CLINICAL TRIAL: NCT00617656
Title: Multicenter Phase III, Randomized Study to Evaluate Treatment Customized According to RAP80 and BRCA1 Assessment in Patients With Advanced Non-small-cell Lung Cancer
Brief Title: Study to Evaluate Treatment Customized According to RAP80 and BRCA1 in Patients With Advanced Lung Carcinoma
Acronym: BREC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No safety reasons. Interim analysis shows that the hypothesis superiority of the experimental arm over the control arm- would not be confirmed.
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECP-BREC; 2007-004278-20 (EudraCT Number)
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer; BRCA1 Mutation
Keywords: Lung Cancer; Chemotherapy; Personalized medicine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cisplatin; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: Control (Active Comparator): Docetaxel 75 mg/m2 and cisplatin 75 mg/m2, both on day 1, every 21 days. Total number of cycles: 6
  Interventions: Drug: Cisplatin, Docetaxel
- B1: Experimental group B1 (Experimental): Low RAP expression and any levels of BRCA1 expression: Gemcitabine 1250 mg/m2, days 1 and 8, and Cisplatin 75 mg/m2, day 1. 21-day cycles. Total number of cycles: 6
  Interventions: Drug: Gemcitabine, Cisplatin
- B2: Experimental group B2 (Experimental): Intermediate or high RAP expression and low or intermediate BRCA1 expression: Docetaxel 75 mg/m2 and Cisplatin 75 mg/m2, both administered on day 1, every 21 days. Total number of cycles: 6
  Interventions: Drug: Docetaxel, Cisplatin
- B3: Experimental group B3 (Experimental): Intermediate or high RAP expression and high BRCA1 expression: Docetaxel 75 mg/m2, day 1. 21-day cycles. Total number of cycles: 6
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Cisplatin, Docetaxel — Docetaxel 75 mg/m2 and cisplatin 75 mg/m2, both on day 1, every 21 days. Total number of cycles: 6
  Other Names: Platinol; Taxotere
  Arms: A: Control
Drug: Gemcitabine, Cisplatin — Gemcitabine 1250 mg/m2, days 1 and 8, and Cisplatin 75 mg/m2, day 1. 21-day cycles. Total number of cycles: 6
  Other Names: Gemzar; Platinol
  Arms: B1: Experimental group B1
Drug: Docetaxel, Cisplatin — Docetaxel 75 mg/m2 and Cisplatin 75 mg/m2, both administered on day 1, every 21 days. Total number of cycles: 6
  Other Names: Taxotere; Platinol
  Arms: B2: Experimental group B2
Drug: Docetaxel — Docetaxel 75 mg/m2, day 1. 21-day cycles. Total number of cycles: 6
  Other Names: Taxotere
  Arms: B3: Experimental group B3

SUMMARY:
Primary objective:

· Progression free survival.

Secondary objectives:

* Assess Overall survival of both treatment groups.
* Assess Tumor response rate using RECIST criteria
* Assess Toxicity profile of patients enrolled in the study.
* Exploratory evaluation of potential genetic markers of response or resistance to chemotherapy.

DETAILED DESCRIPTION:
Study population:

Patients with advanced non-small-cell lung cancer who have not received treatment for the disease at this stage and who have a good performance status (ECOG 0-1) and measurable disease (at least one target lesion according to RECIST criteria).

Duration of treatment:

Six chemotherapy cycles will be given. The duration of every cycle will be 21 days. If the treatment is beneficial, it may be prolonged to a total of 8 cycles at the discretion of the investigator.

Calendar and planned finalization date:

The approximate duration of the study is 3 years of recruitment followed by 1 year of follow-up.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patients age 18 years or more.
2. Histologically confirmed diagnosis of non-small-cell lung carcinoma.
3. Only patients with advanced disease defined as stage IV or IIIB with or without pleural effusion will be included. In the event of IIIB disease without pleural effusion those patients, who for some reason (respiratory disease, large radiation volume...) may not be candidates to have chemotherapy and radiotherapy treatment and may only be treated with chemotherapy, will be considered.
4. Tumor specimen available (according to the criterion of the specimen-processing laboratory) for the analysis of RAP80 and BRCA1 expression in mRNA.
5. A measurable lesion, as defined by RECIST criteria.
6. Karnofsky score 80% or more (ECOG < 2).
7. No previous treatment with chemotherapy or other agents for disseminated disease. Chemotherapy is allowed if the patient's initial diagnosis is limited disease and the patient has received adjuvant or neoadjuvant treatment, as long as a minimum of 6 months has passed since the end of the adjuvant and/or neo-adjuvant chemotherapy.
8. Patients with cerebral disease may be included without any time limitations after holocranial irradiation or complementary antiedema treatment, as long as there is correct control of the clinical symptoms arising from the brain disease or is symptomatic.
9. Patients with the following hematologic values:

   ANC ≥ 1.5 x 109/L Hb ≥ 10 g/dl Platelets ≥ 100 x 109/L
10. Patients with the following biochemical values:

    Bilirubin ≤ 1.5 mg/dL AST and ALT < 1.5 upper limit of normality Creatinine clearance ≥ 60 ml/min.
11. Patients of childbearing age of either sex must use effective contraceptive methods (barrier methods or other birth control methods) before entering the study and while participating in the study.
12. Patients should sign an informed consent form before inclusion in the study that specifies that the clinical trial treatment entails consent for the analysis of biological specimens of tumor and blood.
13. Patients must be available for clinical follow-up.

EXCLUSION CRITERIA

1. Previous chemotherapy treatment, except the supposition reflected in inclusion criterion 7.
2. Patients diagnosed of another neoplasm, with the exception of cervical carcinoma in situ, treated squamous cell carcinomas or superficial bladder tumors (Ta and TIS), or other malignant tumors that have received curative treatment within the last 5 years before inclusion in the study.
3. Patients with serious active bacterial or fungal infective processes from a clinical vantage point (= grade 2 of NCI-CTC, Version 3).
4. Patients who have received an investigational medicinal product in the 21 days before inclusion in the study.
5. Patients with HIV infection, HCV infection, coronary artery disease or uncontrolled arrhythmia, uncontrolled cerebrovascular disease, or other clinical conditions that, in the judgment of the investigator, contraindicate the patient's participation in the study.
6. Patients who are pregnant or breastfeeding. Women of childbearing age must have a negative pregnancy test performed within 7 days before the onset of treatment.
7. Substance abuse and clinical, psychological or social conditions that can undermine the validity of the informed consent or protocol compliance.
8. Patients who present any contraindication or suspected allergy to the products under investigation in the study
9. Impossibility to comply with chemotherapy treatment due to cultural or geographic circumstances.
10. Significant weight loss (= 10% of body weight) in the 6 weeks before inclusion in the study.
11. Any condition that is unstable or could endanger the patient's safety and/or the patient's compliance with the study.
12. Contraindication for steroid use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2008-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafel Rossell, MD, Principal Investigator — Principal Investigator of Fundación Grupo Español de Cáncer de Pulmón
Locations (44):
- Spain (44):
  - H. Virgen de los Lirios, Alcoy, Alicante
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital D'Althaia, Manresa, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital de Cruces, Barakaldo, Bizkaia
  - Hospital Reina Sofía, Córdoba, Córdoba
  - F.H.Alcorcón, Alcorcón, Madrid
  - H. Severo Ochoa, Leganés, Madrid
  - Clinica Quiron, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Ernest Lluch, Calatayud, Zaragoza
  - H. Juan Canalejo, A Coruña
  - H. Santiago de Compostela, A Coruña
  - H. Gral. Alicante, Alicante
  - H. Torrecárdenas, Almería
  - Hospital Torrecárdenas, Almería
  - H. Clinic i Provincial, Barcelona
  - H. Universitario Quirón Dexeus, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - H. Duran i Reynals-ICO, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital General Yagüe, Burgos
  - H. Provincial de Castellón, Castelló
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Ciudad de Jaén, Jaén
  - H. de la Princesa, Madrid
  - H.U. Puerta de Hierro, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Messeguer, Murcia
  - Hospital Son Dureta/ Ses Espases, Palma de Mallorca
  - H. Son Llátzer, Palma de Mallorca
  - Hospital nuestra señora de Valme, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - H. Gen. Univ. Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - H. General de Vic, Vic
  - Hospital Clínico Lozano Blesa, Zaragoza
  - H. Clínico Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karachaliou N, Bracht JWP, Fernandez Bruno M, Drozdowskyj A, Gimenez Capitan A, Moran T, Carcereny E, Cobo M, Domine M, Chaib I, Ramirez JL, Camps C, Provencio M, Vergnenegre A, Lopez-Vivanco G, Majem M, Massuti B, Rosell R. Association of PALB2 Messenger RNA Expression with Platinum-Docetaxel Efficacy in Advanced Non-Small Cell Lung Cancer. J Thorac Oncol. 2019 Feb;14(2):304-310. doi: 10.1016/j.jtho.2018.10.168. Epub 2018 Nov 22. PMID 30472259
- [Derived] Moran T, Wei J, Cobo M, Qian X, Domine M, Zou Z, Bover I, Wang L, Provencio M, Yu L, Chaib I, You C, Massuti B, Song Y, Vergnenegre A, Lu H, Lopez-Vivanco G, Hu W, Robinet G, Yan J, Insa A, Xu X, Majem M, Chen X, de Las Penas R, Karachaliou N, Sala MA, Wu Q, Isla D, Zhou Y, Baize N, Zhang F, Garde J, Germonpre P, Rauh S, ALHusaini H, Sanchez-Ronco M, Drozdowskyj A, Sanchez JJ, Camps C, Liu B, Rosell R; Spanish Lung Cancer Group, the French Lung Cancer Group and the Comprehensive Cancer Centre of Drum Tower Hospital in Nanjing; Colinet B, De Greve J, Germonpre P, Chen H, Chen X, Du J, Gao Y, Hu J, Hu W, Kong W, Li L, Li R, Li X, Liu B, Liu J, Lu H, Qian X, Ren W, Song Y, Wang L, Wei J, Wen L, Wu Q, Xiao X, Xu X, Yan J, Yang J, Yang M, Yang Y, Yin J, You C, Yu L, Yue X, Zhang F, Zhang J, Zhou Y, Zhu L, Zou Z, Baize N, Bombaron P, Chouaid C, Dansin E, Fournel P, Fraboulet G, Gervais R, Hominal S, Kahlout S, Lecaer H, Lena H, LeTreut J, Locher C, Molinier O, Monnet I, Oliviero G, Robinet G, Schoot R, Thomas P, Vergnenegre A, Berchem G, Rauh S, Al Husaini H, Aparisi F, Arriola E, Ballesteros I, Barneto I, Bernabe R, Blasco A, Bosch-Barrera J, Bover I, Calvo de Juan V, Camps C, Carcereny E, Catot S, Cobo M, De Las Penas R, Domine M, Felip E, Garcia-Campelo MR, Garcia-Giron C, Garcia-Gomez R, Garcia-Sevila R, Garde J, Gasco A, Gil J, Gonzalez-Larriba JL, Hernando-Polo S, Jantus E, Insa A, Isla D, Jimenez B, Lianes P, Lopez-Lopez R, Lopez-Martin A, Lopez-Vivanco G, Macias JA, Majem M, Marti-Ciriquian JL, Massuti B, Montoyo R, Morales-Espinosa D, Moran T, Moreno MA, Pallares C, Parera M, Perez-Carrion R, Porta R, Provencio M, Reguart N, Rosell R, Rosillo F, Sala MA, Sanchez JM, Sullivan I, Terrasa J, Trigo JM, Valdivia J, Vinolas N, Viteri S, Botia-Castillo M, Mate JL, Perez-Cano M, Ramirez JL, Sanchez-Rodriguez B, Taron M, Tierno-Garcia M, Mijangos E, Ocana J, Pereira E, Shao J, Sun X, O'Brate R. Two biomarker-directed randomized trials in European and Chinese patients with nonsmall-cell lung cancer: the BRCA1-RAP80 Expression Customization (BREC) studies. Ann Oncol. 2014 Nov;25(11):2147-2155. doi: 10.1093/annonc/mdu389. Epub 2014 Aug 27. PMID 25164908
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There has been a total screening of 1161 patients from which a total of 382 patients could finally be included and randomized.
Groups:
- A Control Group: Docetaxel 75 mg/m2 and cisplatin 75 mg/m2, both on day 1, every 21 days. Total number of cycles: 6
  Cisplatin, Docetaxel: Docetaxel 75 mg/m2 and cisplatin 75 mg/m2, both on day 1, every 21 days. Total number of cycles: 6
- Experimental Group Arm B1: Patients with low expression of RAP 80, and with any level of BRCA1 expression:
  gemcitabine 1250 mg/m2, days 1 and 8, and cisplatin 75 mg/m2, day 1. Cycles every 21 days.
- Experimental Group Arm B2: Patients with intermediate or high expression of RAP 80, and with low or intermediate expression of BRCA1: docetaxel 75 mg/m2, and cisplatin 75 mg/m2, both administered on day 1, every 21 days
- Experimental Group Arm B3: Patients with intermediate or high expression of RAP 80, and with high expression of BRCA1: docetaxel 75 mg/m2, day 1. Cycles every 21 days.
Period: Overall Study
Arm/Group | A Control Group | Experimental Group Arm B1 | Experimental Group Arm B2 | Experimental Group Arm B3
Started | 190 | 81 | 62 | 49
Completed | 142 | 45 | 49 | 43
Not Completed | 48 | 36 | 13 | 6
Not completed — Inclusion error | 4 | 4 | 0 | 0
Not completed — Missing data | 44 | 30 | 13 | 6
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patient valid to intention to treat
Groups:
- Experimental Group: Include experimental groups Arm B1+ Arm B2+ Arm B3
- Total: Total of all reporting groups
Arm/Group | A Control Group | Experimental Group | Total
Number analyzed (Participants) | 142 | 137 | 279
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 82] | 63 [37 to 83] | 62.5 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 19 | 52
  Male | 109 | 118 | 227
Region of Enrollment [Number; unit: participants]
  Spain | 142 | 137 | 279
Smoking status [Number; unit: participants]
  Smoker | 38 | 36 | 74
  Non-smoker | 97 | 95 | 192
  No data | 7 | 6 | 13
ECOG [Number; unit: participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  participants
    ECOG 0 | 44 | 49 | 93
    ECOG 1-2 | 98 | 88 | 186
Stage IV disease extension at study entrance [Number; unit: participants]
  Thoracic | 16 | 12 | 28
  Extra-thoracic | 124 | 123 | 247
  No data | 2 | 2 | 4
Histology [Number; unit: participants]
  Squamous | 50 | 49 | 99
  NonSquamous | 92 | 88 | 180
Median number of cycles [Median (Full Range); unit: cycles] | 5 [1 to 8] | 4 [1 to 7] | 4.5 [1 to 8]
BRCA1 mRNA level [Number; unit: participants] — The expression of BRCA1 mRNA will be determined by RT- PCR in paraffin-embedded tumor samples
  participants
    Low BRCA mRNA level | 50 | 48 | 98
    Intermediate BRCA mRNA level | 46 | 42 | 88
    Hight BRCA mRNA level | 46 | 47 | 93
RAP 80 mRNA level [Number; unit: participants] — The expression of RAP80 mRNA will be determined by RT-PCR in paraffin-embedded tumor samples
  participants
    Low RAP80 mRNA level | 52 | 48 | 100
    Intermediate RAP80 mRNA level | 50 | 55 | 105
    Hight RAP80 mRNA level | 36 | 34 | 70
    Undetermined level RAP80 mRNA | 4 | 0 | 4
mRNA RAP80 expression values [Median (Full Range); unit: fg/μg] — mRNA expression by a real-time PCR in paraffin-embedded tumor samples
  fg/μg | 1.65 [0.33 to 16.91] | 1.74 [0.32 to 10.19] | 1.7 [0.32 to 16.91]
mRNA BRCA1 expression values [Median (Full Range); unit: fg/μg] — mRNA expression by a real-time PCR in paraffin-embedded tumor samples
  fg/μg | 11.86 [0.49 to 149.53] | 12.28 [0.77 to 48.06] | 12 [0.49 to 149.53]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Defined as the length of time from the start of treatment to the date of the first documented progression of disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the day of start of treatment until first documented progression or death due to any cause,up to 18 months.
Measure: Median (95% Confidence Interval); unit: Month
Groups:
- Control Group: Docetaxel 75 mg/m2 and cisplatin 75 mg/m2, both on day 1, every 21 days. Total number of cycles: 6
  Cisplatin, Docetaxel: Docetaxel 75 mg/m2 and cisplatin 75 mg/m2, both on day 1, every 21 days. Total number of cycles: 6
- B1: Experimental Group 1: Low RAP expression and any levels of BRCA1 expression: Gemcitabine 1250 mg/m2, days 1 and 8, and Cisplatin 75 mg/m2, day 1. 21-day cycles. Total number of cycles: 6
  Gemcitabine, Cisplatin: Gemcitabine 1250 mg/m2, days 1 and 8, and Cisplatin 75 mg/m2, day 1. 21-day cycles. Total number of cycles: 6
- B2 Experimental Group 2: Intermediate or high RAP expression and low or intermediate BRCA1 expression: Docetaxel 75 mg/m2 and Cisplatin 75 mg/m2, both administered on day 1, every 21 days. Total number of cycles: 6
  Docetaxel, Cisplatin: Docetaxel 75 mg/m2 and Cisplatin 75 mg/m2, both administered on day 1, every 21 days. Total number of cycles: 6
- B3 Experimental Group 3: Intermediate or high RAP expression and high BRCA1 expression: Docetaxel 75 mg/m2, day 1. 21-day cycles. Total number of cycles: 6
  Docetaxel: Docetaxel 75 mg/m2, day 1. 21-day cycles. Total number of cycles: 6
Arm/Group | Control Group | B1: Experimental Group 1 | B2 Experimental Group 2 | B3 Experimental Group 3
Number analyzed (Participants) | 142 | 45 | 49 | 43
Month | 5.49 [5.08 to 5.91] | 5.43 [5.08 to 5.77] | 5.49 [3.83 to 7.16] | 2.50 [1.16 to 3.84]
Statistical Analysis 1: Comparison: Control Group vs B1: Experimental Group 1; This is a futility analysis. The initial hypothesis of the clinical trial was that the experimental group as a whole was superior to the control group; Test type: Superiority; p = 0.56, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.76 to 1.67]
Statistical Analysis 2: Comparison: Control Group vs B2 Experimental Group 2; Test type: Superiority; p = 0.79, Log Rank; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.73 to 1.51]
Statistical Analysis 3: Comparison: Control Group vs B3 Experimental Group 3; Test type: Superiority; p = 0.0001, Log Rank; Hazard Ratio (HR) = 2.02, 95% CI 2-sided [1.38 to 2.95]

2. Secondary Outcome: Overall Survival
Description: Defined as the length of time from the start of the treatment that patients diagnosed with the disease are still alive.
Time Frame: From the date of start of the treatment until death or end of follow up, up to 18 months.
Measure: Median (95% Confidence Interval); unit: Month
Groups:
- Experimental Group: Include experimental groups 1, 2 & 3
Arm/Group | A Control Group | Experimental Group
Number analyzed (Participants) | 142 | 137
Month | 12.66 [10.07 to 15.26] | 8.52 [6.41 to 10.63]
Statistical Analysis 1: Comparison: A Control Group vs Experimental Group; Test type: Superiority; p = 0.006, Log Rank; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [1.13 to 2.12]

ADVERSE EVENTS:
Time Frame: 60 Months
Description: The drugs used in this trial have been on the market for several years and the profile of safety is known. No unusual AEs has occurred in this trial.
  Since the objective of the interim analysis for which the trial was closed was not the analysis of AEs, these have not been analyzed for this trial.
  During the study were reported 68 cases of SAEs related to medication and 106 cases of SAEs not related to medication.
  The only SUSAR was: Severe afebrile neutropenia and renal failure.
Arm/Group | Control Group | B1: Experimental Group 1 | B2 Experimental Group 2 | B3 Experimental Group 3
All-Cause Mortality (participants affected / at risk) | 2/142 | 7/45 | 19/49 | 3/43
Serious Adverse Events (participants affected / at risk) | 9/142 | 29/45 | 49/49 | 6/43
Other Adverse Events (participants affected / at risk) | 0/142 | 0/45 | 0/49 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=142) | B1: Experimental Group 1 (N=45) | B2 Experimental Group 2 (N=49) | B3 Experimental Group 3 (N=43)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 24 (24) | 1 (1)
Tromboembolismo pulmonar (Vascular disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 5 (5) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 5 (5) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 5 (5) | 3 (3) | 1 (1)
Asthenia (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Confusional syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumoniae (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 8 (8) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The were a early closure of the study and it was notified to comply with the regulations for early termination of the studies. clinical trials (futility analysis).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No